CLINICAL TRIAL: NCT04381650
Title: A Phase 1b/2 Study of TAK-981 Plus Pembrolizumab to Evaluate the Safety, Tolerability, and Antitumor Activity of the Combination in Patients With Select Advanced or Metastatic Solid Tumors
Brief Title: A Study of TAK-981 Given With Pembrolizumab in Participants With Select Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TAK-981-1502; 2020-004325-23 (EudraCT Number); jRCT2031210417 (Registry Identifier: jRCT)
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Results first posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Advanced or Metastatic Solid Tumors
Keywords: Drug Therapy
MeSH Terms: interventions — TAK-981; pembrolizumab

STUDY DESIGN:
Intervention Model Description: This study has 2 Phases. Phase 1 is dose escalation phase with sequential drug assignment. Phase 2 is parallel assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (11):
- Dose Escalation: TAK-981 40 mg + Pembrolizumab (Experimental): Participants received TAK-981 40 mg, intravenous (IV) infusion, on Days 1, 4, 8 and 11 or Days 1 and 8 in each 21-day Treatment Cycle and pembrolizumab 200 mg, IV infusion, as a fixed dose every 3 weeks on Day 1 of 21-day Treatment Cycle until the recommended Phase 2 dose (RP2D) was determined (for a maximum of 24 months).
  Interventions: Drug: TAK-981; Drug: Pembrolizumab
- Dose Escalation: TAK-981 60 mg + Pembrolizumab (Experimental): Participants received TAK-981 60 mg, intravenous (IV) infusion, on Days 1, 4, 8 and 11 or Days 1 and 8 in each 21-day Treatment Cycle and pembrolizumab 200 mg, IV infusion, as a fixed dose every 3 weeks on Day 1 of 21-day Treatment Cycle until the RP2D was determined (for a maximum of 24 months).
  Interventions: Drug: TAK-981; Drug: Pembrolizumab
- Dose Escalation: TAK-981 90 mg + Pembrolizumab (Experimental): Participants received TAK-981 90 mg, intravenous (IV) infusion, on Days 1, 4, 8 and 11 or Days 1 and 8 in each 21-day Treatment Cycle and pembrolizumab 200 mg, IV infusion, as a fixed dose every 3 weeks on Day 1 of 21-day Treatment Cycle until the RP2D was determined (for a maximum of 24 months).
  Interventions: Drug: TAK-981; Drug: Pembrolizumab
- Dose Escalation: TAK-981 120 mg + Pembrolizumab (Experimental): Participants received TAK-981 120 mg, intravenous (IV) infusion, on Days 1, 4, 8 and 11 or Days 1 and 8 in each 21-day Treatment Cycle and pembrolizumab 200 mg, IV infusion, as a fixed dose every 3 weeks on Day 1 of 21-day Treatment Cycle until the RP2D was determined (for a maximum of 24 months).
  Interventions: Drug: TAK-981; Drug: Pembrolizumab
- Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 90 mg (Experimental): Participants with non-squamous non-small cell lung cancer (NSCLC) received TAK-981 as IV infusion on Days 1, 4, 8 and 11 or Days 1 and 8 in each 21-day Treatment Cycle up to disease progression or 24-months and pembrolizumab 200 mg IV infusion as a fixed dose every 3 weeks on Day 1 of 21-day Treatment Cycle for a maximum of 24 months.
  Interventions: Drug: TAK-981; Drug: Pembrolizumab
- Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 120 mg (Experimental): Participants with NSCLC received TAK-981 as IV infusion on Days 1, 4, 8 and 11 or Days 1 and 8 in each 21-day Treatment Cycle up to disease progression or 24-months and pembrolizumab 200 mg IV infusion as a fixed dose every 3 weeks on Day 1 of 21-day Treatment Cycle for a maximum of 24 months.
  Interventions: Drug: TAK-981; Drug: Pembrolizumab
- Dose Expansion Phase: Cohort B: Cervical Cancer (Experimental): Participants with cervical cancer received TAK-981 as IV infusion on Days 1, 4, 8 and 11 or Days 1 and 8 in each 21-day Treatment Cycle up to disease progression or 24-months and pembrolizumab 200 mg IV infusion as a fixed dose every 3 weeks on Day 1 of 21-day Treatment Cycle for a maximum of 24 months.
  Interventions: Drug: TAK-981; Drug: Pembrolizumab
- Dose Expansion Phase: Cohort C: MSS-CRC (Experimental): Participants with microsatellite stable colorectal cancer (MSS-CRC) received TAK-981 as IV infusion on Days 1, 4, 8 and 11 or Days 1 and 8 in each 21-day Treatment Cycle up to disease progression or 24-months and pembrolizumab 200 mg IV infusion as a fixed dose every 3 weeks on Day 1 of 21-day Treatment Cycle for a maximum of 24 months.
  Interventions: Drug: TAK-981; Drug: Pembrolizumab
- Dose Expansion Phase: Cohort D: Cutaneous Melanoma (Experimental): Participants with cutaneous melanoma received TAK-981 as IV infusion on Days 1, 4, 8 and 11 or Days 1 and 8 in each 21-day Treatment Cycle up to disease progression or 24-months and pembrolizumab 200 mg IV infusion as a fixed dose every 3 weeks on Day 1 of 21-day Treatment Cycle for a maximum of 24 months.
  Interventions: Drug: TAK-981; Drug: Pembrolizumab
- Dose Expansion Phase: Cohort E: Squamous NSCLC (Experimental): Participants with squamous NSCLC received TAK-981 as IV infusion on Days 1, 4, 8 and 11 or Days 1 and 8 in each 21-day Treatment Cycle up to disease progression or 24-months and pembrolizumab 200 mg IV infusion as a fixed dose every 3 weeks on Day 1 of 21-day Treatment Cycle for a maximum of 24 months.
  Interventions: Drug: TAK-981; Drug: Pembrolizumab
- Dose Expansion Phase: Cohort F: CPI Refractory Squamous or Nonsquamous NSCLC (Experimental): Participants with checkpoint inhibitors (CPI) refractory squamous or non-squamous NSCLC received TAK-981 as IV infusion on Days 1, 4, 8 and 11 or Days 1 and 8 in each 21-day Treatment Cycle up to disease progression or 24-months and pembrolizumab 200 mg IV infusion as a fixed dose every 3 weeks on Day 1 of 21-day Treatment Cycle for a maximum of 24 months.
  Interventions: Drug: TAK-981; Drug: Pembrolizumab

INTERVENTIONS:
Drug: TAK-981 — TAK-981 IV infusion.
Drug: Pembrolizumab — Pembrolizumab IV infusion.

SUMMARY:
TAK-981 is being tested in combination with pembrolizumab to treat participants who have select advanced or metastatic solid tumors.

The study aims are to evaluate the safety, tolerability, and preliminary efficacy of TAK-981 in combination with pembrolizumab.

Participants will be on this combination treatment for 21-day cycles. They will continue with this treatment for up to 24 months or until participants meet any discontinuation criteria.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-981. TAK-981 is being tested to treat people who have select advanced or metastatic solid tumors. The study will include a dose escalation phase and a dose expansion phase.

The study will enroll approximately 231 participants, approximately 32 participants in the dose escalation phase 1 and approximately 76 to 199 participants in the 8 cohorts of dose expansion phase 2. Participants will receive escalating doses of TAK-981 and fixed dose of pembrolizumab until recommended phase 2 dose (RP2D) is determined:

• Dose Escalation: TAK-981 + Pembrolizumab (Fixed Dose)

Once Phase 2 doses are identified, participants of select advanced or metastatic solid tumors will receive TAK-981 in below defined cohorts in the expansion phase 2:

* Dose Expansion Phase: Cohort A: Non-squamous Non-small Cell Lung Cancer (NSCLC)
* Dose Expansion Phase: Cohort B: Cervical Cancer
* Dose Expansion Phase: Cohort C: Microsatellite Stable Colorectal Cancer (MSS-CRC)
* Dose Expansion Phase: Cohort D: Cutaneous Melanoma
* Dose Expansion Phase: Cohort E: Squamous NSCLC
* Dose Expansion Phase: Cohort F: Checkpoint Inhibitors (CPI) Refractory Squamous or Nonsquamous NSCLC

This multi-center trial will be conducted worldwide. The overall time to participate in this study is 60 months. Participants will make multiple visits to the clinic, and progression-free survival follow-up for maximum up to 12 months after last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Has a histologically or cytologically documented, advanced (metastatic and/or unresectable) cancer as listed below that is incurable: Note: Prior neoadjuvant or adjuvant therapy included in initial treatment may not be considered first- or later-line standard of care treatment unless such treatments were completed less than 12 months prior to the current tumor recurrence.

   A. Non-squamous NSCLC for which prior standard first-line treatment containing an anti-programmed cell death protein 1/programmed cell death protein 1 ligand (PD-1/PD-L1) checkpoint inhibitor (CPI) alone or in combination has failed and that has progressed on no more than 1 prior systemic therapy. In Phase 2, participants with nonsquamous NSCLC must have not received more than 1 prior systemic therapy and must not have presented with disease progression during the first 6 months of treatment with first-line CPI/anti-PD-(1/L1)-containing therapy.

   Note: In Phase 1, participants with nonsquamous NSCLC and known driver mutations/genomic aberrations (e.g., epidermal growth factor receptor (EGFR), B-Raf proto-oncogene mutation V600E [BRAF V600E], and ROS proto-oncogene 1 [ROS1] sensitizing mutations, neurotrophic receptor tyrosine kinase [NRTK] gene fusions, and anaplastic lymphoma kinase [ALK] rearrangements) must have also shown progressive disease after treatment with a commercially available targeted therapy. In Phase 2, participants with driver mutations are not eligible.

   B. CPI-naive cervical cancer (squamous cell carcinoma, adenosquamous carcinoma or adenocarcinoma of the cervix) participants for whom prior standard first-line treatment has failed and who have received no more than 1 prior systemic line of therapy for recurrent or Stage IVB cervical cancer. Note: The following cervical tumors are not eligible: minimal deviation/adenoma malignum, gastric-type adenocarcinoma, clear-cell carcinoma, and mesonephric carcinoma. Histologic confirmation of the original primary tumor is required via pathology report. Note: First-line treatment must have consisted of platinum-containing doublet. Chemotherapy administered concurrently with primary radiation (e.g., weekly cisplatin) is not counted as a systemic chemotherapy regimen.

   C. CPI-naïve microsatellite stable-colorectal cancer (MSS-CRC) participants for whom prior standard first-line treatment has failed and who have progressed on no more than 3 chemotherapy regimens.

   Note: Participants must have received prior treatment with fluoropyrimidine-, oxaliplatin-, and irinotecan-containing regimens if indicated.

   D. Unresectable Stage III or Stage IV cutaneous melanoma that has not received prior therapy in the metastatic setting.

   Note: Participants with acral melanoma are not eligible. Participants who have presented with disease relapse after ≥6 months of the last dose of CPI or BRAF-mitogen-activated protein kinase kinase (MEK) inhibitor in the adjuvant setting are eligible.

   E. Squamous NSCLC for which prior standard first-line treatment containing an anti-PD-(1/L1) checkpoint inhibitor alone or in combination has failed. Participant must have not received more than 1 prior systemic therapy and must not have presented with disease progression during the first 6 months of treatment with first-line CPI/anti-PD-(1/L1)-containing therapy.

   F. Squamous or nonsquamous NSCLC for which prior standard first-line treatment containing an anti-PD-(1/L1) checkpoint inhibitor alone or in combination has failed within 6 months from the initiation of the CPI. Participants must not have received more than 1 prior systemic therapy in the metastatic setting.

   Note: Participants with driver mutations are not eligible.
2. Has at least 1 radiologically measurable lesion based on RECIST, Version 1.1. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
3. Has a performance status of 0 or 1 on the Eastern Cooperative Group Oncology (ECOG) Performance Scale.
4. Has left ventricular ejection fraction (LVEF) ≥40%; as measured by echocardiogram (ECHO) or multiple-gated acquisition (MUGA) scan.
5. Has recovered to Grade 1 or baseline from all toxicity associated with previous therapy or have the toxicity established as sequela. Note: Has a neuropathy ≤Grade 2, any grade alopecia, or autoimmune endocrinopathies with stable replacement therapy are permitted.
6. Demonstrate adequate organ function as described below:

A. Platelet count ≥75.0 × 10^9/L. B. Absolute neutrophil count (ANC) ≥1.0 × 10^9/L. C. Hemoglobin ≥85 g/L (red blood cell [RBC] transfusion allowed ≥14 days before assessment).

D. Calculated creatinine clearance ≥30 mL/min using the Cockcroft-Gault formula.

E. Aspartate aminotransferase (AST, GOT) and alanine aminotransferase (ALT, GPT) ≤3.0 times the upper limit of normal (ULN), <5.0 times the ULN if liver enzyme elevations are due to liver metastases; bilirubin ≤1.5 times the ULN. Participants with Gilbert's syndrome may have a bilirubin level >1.5 times the ULN, per discussion between the investigator and the medical monitor.

Exclusion Criteria:

1. History of uncontrolled brain metastasis (evidence of progression by imaging over a period of 4 weeks and/or neurologic symptoms that have not returned to baseline). Participant with treated brain metastases are allowed provided they are radiologically stable, without evidence of progression for at least 4 weeks by repeat imaging, clinically stable, and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment. Note: For asymptomatic participants, screening brain imaging is not required.
2. Second malignancy within the previous 3 years, except treated basal cell or localized squamous skin carcinomas, localized prostate cancer, cervical carcinoma in situ, resected colorectal adenomatous polyps, breast cancer in situ, or other malignancy for which the participant is not on active anticancer therapy.
3. Major surgery ≤14 days from the first dose of study drug and not recovered fully from any complications from surgery.
4. History of immune-related AEs related to treatment with immune CPIs that required treatment discontinuation.
5. Receiving or requires the continued use of medications that are known to be strong or moderate inhibitors and inducers of cytochrome P-450 (CYP) 3A4/5 and strong P-glycoprotein (Pgp) inhibitors.
6. Baseline prolongation of the QT interval corrected using Fridericia's formula (QTcF) (e.g., repeated demonstration of QTcF interval >480 milliseconds (ms), history of congenital long QT syndrome, or torsades de pointes).
7. Has a history of autoimmune disease requiring systemic immunosuppressive therapy with daily doses of prednisone >10 mg/day or equivalent doses, or any other form of immunosuppressive therapy. Hormone replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for thyroid, adrenal or pituitary insufficiency) for endocrinopathies are not considered prohibited forms of systemic treatment of an autoimmune disease.
8. Has a history of noninfectious pneumonitis that required steroids or a history of interstitial lung disease.
9. Has an evidence of active, non-infectious pneumonitis.
10. Has a history of allogeneic tissue or solid organ transplant.
11. Has an active infection requiring systemic therapy.
12. Has a known history of human immunodeficiency virus (HIV) infection or any other relevant congenital or acquired immunodeficiency.
13. Has a known hepatitis B virus surface antigen seropositive or detectable hepatitis C infection viral load. Note: Participants who have positive hepatitis B core antibody or hepatitis B surface antigen antibody can be enrolled but must have an undetectable hepatitis B viral load.
14. History of any of the following ≤6 months before first dose: congestive heart failure New York Heart Association Grade III or IV, unstable angina, myocardial infarction, unstable symptomatic ischemic heart disease, uncontrolled hypertension despite appropriate medical therapy, ongoing symptomatic cardiac arrhythmias >Grade 2, pulmonary embolism or symptomatic cerebrovascular events, or any other serious cardiac condition (e.g., pericardial effusion or restrictive cardiomyopathy). Chronic atrial fibrillation on stable anticoagulant therapy is allowed.
15. Psychiatric illness/social circumstances that would limit compliance with study requirements and substantially increase the risk of AEs or has compromised ability to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (52):
- United States (18):
  - HonorHealth, Scottsdale, Arizona
  - University of California Irvine Medical Center, Orange, California
  - Stanford Cancer Institute (SCI), Stanford, California
  - Yale Cancer Center, New Haven, Connecticut
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - The Center for Cancer and Blood Disorders - PPDS, Bethesda, Maryland
  - Morristown Medical Center, Morristown, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Montefiore Einstein Cancer Center - BRANY - PPDS, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Oklahoma Peggy and Charles Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Providence Cancer Institute, Franz Clinic, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - START South Texas Accelerated Research Therapeutics, San Antonio, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Virginia Cancer Specialists (Fairfax) - USOR, Fairfax, Virginia
- Brazil (9):
  - Instituto de Oncologia Do Parana, Curitiba, Paraná
  - ONCOSITE Centro de Pesquisa Clinica Em Oncologia, Ijuí, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre (HCPA) - PPDS, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas Da Pontificia Universidade Catolica Do Rio Grande Do Sul (PUCRS), Porto Alegre, Rio Grande do Sul
  - Fundacao Pio XII Hospital de Cancer de Barretos, Barretos, São Paulo
  - Hospital de Base Da Faculdade de Medicina de Sao Jose Do Rio Preto, São José do Rio Preto, São Paulo
  - Cetus Hospital Dia Oncologia, Belo Horizonte
  - INCA Instituto Nacional de Cancer, Rio de Janeiro
  - Instituto Do Cancer Do Estado de Sao Paulo Octavio Frias de Oliveira, Rio de Janeiro
- China (3):
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Affiliated Hospital, Zhejiang University School of Medicine - PPDS, Hangzhou, Zhejiang
- Croatia (4):
  - Klinicki bolnicki centar Zagreb, Zagreb, City of Zagreb
  - Clinical Hospital Centre Osijek, Osijek
  - General Hospital Pula, Pula
  - University Hospital Centre Split, Split
- Japan (3):
  - National Cancer Center East, Kashiwa-Shi, Chiba
  - National Cancer Center Hospital, Chuo-Ku, Tokyo
  - The Cancer Institute Hospital of Japanese Foundation For Cancer Research, Chuo-Ku, Tokyo
- Latvia (2):
  - Pauls Stradins Clinical University Hospital, Riga
  - Riga East Clinical University Hospital Latvian Oncology Center, Riga
- Lithuania (3):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas, Kaunas County
  - Hospital of Lithuanian University of Health Sciences Kauno klinikos, Kaunas, Kaunas County
  - National Cancer Institute, Vilnius, Vilnius County
- Poland (7):
  - Uniwersyteckie Centrum Kliniczne-Ul. Smoluchowskiego 17, Gdansk, Pomeranian Voivodeship
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka w Bydgoszczy, Bydgoszcz
  - Instytut Medyczny Santa Familia Sp. z o. o., Lodz
  - Specjalistyczna Praktyka Lekarska Slawomir Mandziuk, Lublin
  - Warminsko-Mazurskie Centrum Chorob Pluc w Olsztynie, Olsztyn
  - Med-Polonia Sp. z o.o., Poznan
  - Centrum Terapii Wspolczesnej, Lodz, Łódź Voivodeship
- Switzerland (3):
  - Kantonsspital Muensterlingen, Münsterlingen, Thurgau (de)
  - Kantonsspital Winterthur, Winterthur, Zurich (de)
  - Universitaetsspital Bern - Inselspital, Bern

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Nakamura A, Grossman S, Song K, Xega K, Zhang Y, Cvet D, Berger A, Shapiro G, Huszar D. The SUMOylation inhibitor subasumstat potentiates rituximab activity by IFN1-dependent macrophage and NK cell stimulation. Blood. 2022 May 5;139(18):2770-2781. doi: 10.1182/blood.2021014267. PMID 35226739
- See also: To obtain more information about this study, click this link. — https://clinicaltrials.takeda.com/study-detail/5f6b603d4db2bf003ab4a3a5?idFilter=%5B%22TAK-981-1502%22%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at various investigative sites throughout the world from 17 August 2020 to 29 October 2024.
Pre-assignment Details: Participants with a diagnosis of advanced or metastatic solid tumors were enrolled in this study consisting of Phase 1b (Dose Escalation cohorts), and Phase 2 (Dose Expansion cohorts) periods to receive TAK-981 and pembrolizumab.
Groups:
- Dose Escalation: TAK-981 40 mg: Participants received TAK-981 40 mg, intravenous (IV) infusion, on Days 1, 4, 8 and 11 or Days 1 and 8 in each 21-day Treatment Cycle and pembrolizumab 200 mg, IV infusion, as a fixed dose every 3 weeks on Day 1 of 21-day Treatment Cycle until the recommended Phase 2 dose (RP2D) was determined (for a maximum of 24 months).
- Dose Escalation: TAK-981 60 mg: Participants received TAK-981 60 mg, IV infusion, on Days 1, 4, 8 and 11 or Days 1 and 8 in each 21-day Treatment Cycle and pembrolizumab 200 mg, IV infusion, as a fixed dose every 3 weeks on Day 1 of 21-day Treatment Cycle until the RP2D was determined (for a maximum of 24 months).
- Dose Escalation: TAK-981 90 mg: Participants received TAK-981 90 mg, IV infusion, on Days 1, 4, 8 and 11 or Days 1 and 8 in each 21-day Treatment Cycle and pembrolizumab 200 mg, IV infusion, as a fixed dose every 3 weeks on Day 1 of 21-day Treatment Cycle until the RP2D was determined (for a maximum of 24 months).
- Dose Escalation: TAK-981 120 mg: Participants received TAK-981 120 mg, IV infusion, on Days 1, 4, 8 and 11 or Days 1 and 8 in each 21-day Treatment Cycle and pembrolizumab 200 mg, IV infusion, as a fixed dose every 3 weeks on Day 1 of 21-day Treatment Cycle until the RP2D was determined (for a maximum of 24 months).
- Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 90 mg: Participants with non-squamous non-small cell lung cancer (NSCLC) received TAK-981 90 mg as IV infusion on Days 1, 4, 8 and 11 or Days 1 and 8 in each 21-day Treatment Cycle up to disease progression or 24-months and pembrolizumab 200 mg IV infusion as a fixed dose every 3 weeks on Day 1 of 21-day Treatment Cycle for a maximum of 24 months.
- Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 120 mg: Participants with non-squamous NSCLC received TAK-981 120 mg as IV infusion on Days 1 and 8 in each 21-day Treatment Cycle up to disease progression or 24-months and pembrolizumab 200 mg IV infusion as a fixed dose every 3 weeks on Day 1 of 21-day Treatment Cycle for a maximum of 24 months.
- Dose Expansion: Cohort B: Cervical Cancer TAK-981 90 mg: Participants with cervical cancer received TAK-981 90 mg as IV infusion on Days 1, 4, 8 and 11 or Days 1 and 8 in each 21-day Treatment Cycle up to disease progression or 24-months and pembrolizumab 200 mg IV infusion as a fixed dose every 3 weeks on Day 1 of 21-day Treatment Cycle for a maximum of 24 months.
- Dose Expansion: Cohort C: MSS-CRC TAK-981 90 mg: Participants with microsatellite stable colorectal cancer (MSS-CRC) received TAK-981 90 mg as IV infusion on Days 1, 4, 8 and 11 or Days 1 and 8 in each 21-day Treatment Cycle up to disease progression or 24-months and pembrolizumab 200 mg IV infusion as a fixed dose every 3 weeks on Day 1 of 21-day Treatment Cycle for a maximum of 24 months.
- Dose Expansion: Cohort D: Cutaneous Melanoma TAK-981 90 mg: Participants with cutaneous melanoma received TAK-981 90 mg as IV infusion on Days 1, 4, 8 and 11 or Days 1 and 8 in each 21-day Treatment Cycle up to disease progression or 24-months and pembrolizumab 200 mg IV infusion as a fixed dose every 3 weeks on Day 1 of 21-day Treatment Cycle for a maximum of 24 months.
- Dose Expansion: Cohort E: Squamous NSCLC TAK-981 90 mg: Participants with squamous NSCLC received TAK-981 90 mg as IV infusion on Days 1, 4, 8 and 11 or Days 1 and 8 in each 21-day Treatment Cycle up to disease progression or 24-months and pembrolizumab 200 mg IV infusion as a fixed dose every 3 weeks on Day 1 of 21-day Treatment Cycle for a maximum of 24 months.
- Dose Expansion: Cohort F: CPI Refractory Squamous and Non-squamous NSCLC TAK-981 90 mg: Participants with checkpoint inhibitors (CPI) refractory squamous and non-squamous NSCLC received TAK-981 90 mg as IV infusion on Days 1, 4, 8 and 11 or Days 1 and 8 in each 21-day Treatment Cycle up to disease progression or 24-months and pembrolizumab 200 mg IV infusion as a fixed dose every 3 weeks on Day 1 of 21-day Treatment Cycle for a maximum of 24 months.
Period: Phase 1b (Dose Escalation)
Arm/Group | Dose Escalation: TAK-981 40 mg | Dose Escalation: TAK-981 60 mg | Dose Escalation: TAK-981 90 mg | Dose Escalation: TAK-981 120 mg | Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 90 mg | Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 120 mg | Dose Expansion: Cohort B: Cervical Cancer TAK-981 90 mg | Dose Expansion: Cohort C: MSS-CRC TAK-981 90 mg | Dose Expansion: Cohort D: Cutaneous Melanoma TAK-981 90 mg | Dose Expansion: Cohort E: Squamous NSCLC TAK-981 90 mg | Dose Expansion: Cohort F: CPI Refractory Squamous and Non-squamous NSCLC TAK-981 90 mg
Started | 3 | 6 | 33 | 19 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed (The end of study status for study terminated by sponsor or Death participant is considered as Completed.) | 2 | 2 | 9 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 4 | 24 | 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — New anti-cancer therapy | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 1 | 3 | 12 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 11 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Reason Not Specified | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 2 (Dose Expansion)
Arm/Group | Dose Escalation: TAK-981 40 mg | Dose Escalation: TAK-981 60 mg | Dose Escalation: TAK-981 90 mg | Dose Escalation: TAK-981 120 mg | Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 90 mg | Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 120 mg | Dose Expansion: Cohort B: Cervical Cancer TAK-981 90 mg | Dose Expansion: Cohort C: MSS-CRC TAK-981 90 mg | Dose Expansion: Cohort D: Cutaneous Melanoma TAK-981 90 mg | Dose Expansion: Cohort E: Squamous NSCLC TAK-981 90 mg | Dose Expansion: Cohort F: CPI Refractory Squamous and Non-squamous NSCLC TAK-981 90 mg
Started | 0 | 0 | 0 | 0 | 14 | 9 | 21 | 9 | 28 | 15 | 4
Completed (The end of study status for study terminated by sponsor or Death participant is considered as Completed.) | 0 | 0 | 0 | 0 | 8 | 5 | 17 | 2 | 23 | 4 | 1
Not Completed | 0 | 0 | 0 | 0 | 6 | 4 | 4 | 7 | 5 | 11 | 3
Not completed — New anti-cancer therapy | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 3 | 3 | 4 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 2 | 4 | 2 | 1 | 4 | 1
Not completed — Reason Not Specified | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included participants who received at least 1 dose, even if incomplete, of study drug.
Groups:
- Dose Escalation: TAK-981 40 mg: Participants received TAK-981 40 mg, IV infusion, on Days 1, 4, 8 and 11 or Days 1 and 8 in each 21-day Treatment Cycle and pembrolizumab 200 mg, IV infusion, as a fixed dose every 3 weeks on Day 1 of 21-day Treatment Cycle until the RP2D was determined (for a maximum of 24 months).
- Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 90 mg: Participants with non-squamous NSCLC received TAK-981 90 mg as IV infusion on Days 1, 4, 8 and 11 or Days 1 and 8 in each 21-day Treatment Cycle up to disease progression or 24-months and pembrolizumab 200 mg IV infusion as a fixed dose every 3 weeks on Day 1 of 21-day Treatment Cycle for a maximum of 24 months.
- Dose Expansion: Cohort C: MSS-CRC TAK-981 90 mg: Participants with MSS-CRC received TAK-981 90 mg as IV infusion on Days 1, 4, 8 and 11 or Days 1 and 8 in each 21-day Treatment Cycle up to disease progression or 24-months and pembrolizumab 200 mg IV infusion as a fixed dose every 3 weeks on Day 1 of 21-day Treatment Cycle for a maximum of 24 months.
- Dose Expansion: Cohort F: CPI Refractory Squamous and Non-squamous NSCLC TAK-981 90 mg: Participants with CPI refractory squamous and non-squamous NSCLC received TAK-981 90 mg as IV infusion on Days 1, 4, 8 and 11 or Days 1 and 8 in each 21-day Treatment Cycle up to disease progression or 24-months and pembrolizumab 200 mg IV infusion as a fixed dose every 3 weeks on Day 1 of 21-day Treatment Cycle for a maximum of 24 months.
- Total: Total of all reporting groups
Arm/Group | Dose Escalation: TAK-981 40 mg | Dose Escalation: TAK-981 60 mg | Dose Escalation: TAK-981 90 mg | Dose Escalation: TAK-981 120 mg | Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 90 mg | Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 120 mg | Dose Expansion: Cohort B: Cervical Cancer TAK-981 90 mg | Dose Expansion: Cohort C: MSS-CRC TAK-981 90 mg | Dose Expansion: Cohort D: Cutaneous Melanoma TAK-981 90 mg | Dose Expansion: Cohort E: Squamous NSCLC TAK-981 90 mg | Dose Expansion: Cohort F: CPI Refractory Squamous and Non-squamous NSCLC TAK-981 90 mg | Total
Number analyzed (Participants) | 3 | 6 | 33 | 19 | 14 | 9 | 21 | 9 | 28 | 15 | 4 | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (5.57) | 53.5 (7.23) | 56.2 (11.91) | 59.8 (13.32) | 63.3 (10.83) | 68.7 (9.12) | 51.8 (13.24) | 49.6 (9.22) | 55.9 (13.95) | 67.5 (7.66) | 73.5 (3.70) | 58.5 (12.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 16 | 8 | 6 | 5 | 21 | 5 | 12 | 1 | 1 | 81
  Male | 2 | 1 | 17 | 11 | 8 | 4 | 0 | 4 | 16 | 14 | 3 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 6 | 1 | 5 | 0 | 12 | 0 | 14 | 0 | 0 | 41
  Not Hispanic or Latino | 1 | 5 | 25 | 18 | 8 | 9 | 9 | 9 | 14 | 14 | 4 | 116
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 4 | 8 | 7 | 3 | 1 | 2 | 1 | 4 | 5 | 0 | 35
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 6
  White | 3 | 2 | 17 | 9 | 10 | 8 | 17 | 7 | 23 | 10 | 4 | 110
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 5 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 8

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With One or More Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant administered a medicinal investigational drug. The untoward medical occurrence does not necessarily have to have a causal relationship with treatment. A TEAE is defined as an AE that occurs after administration of first dose of study drug and through 30 days after last dose of study drug or until start of subsequent antineoplastic therapy. AEs were evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 5.0 except cytokine release syndrome (CRS), which was graded according to American Society for Transplantation and Cellular Therapy (ASTCT) Consensus Grading for CRS.
Time Frame: Up to approximately 24 months
Population: Safety Analysis Set included participants who received at least 1 dose, even if incomplete, of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: TAK-981 40 mg | Dose Escalation: TAK-981 60 mg | Dose Escalation: TAK-981 90 mg | Dose Escalation: TAK-981 120 mg
Number analyzed (Participants) | 3 | 6 | 33 | 19
Participants | 3 | 6 | 33 | 19

2. Primary Outcome: Phase 1: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLTs were evaluated according to NCI CTCAE Version 5.0 except CRS, which was graded according to ASTCT Consensus Grading for CRS.
Time Frame: Up to Cycle 1 (each cycle was of 21 days)
Population: The DLT-evaluable Analysis Set included participants enrolled in Phase 1b of the study and who experienced a DLT at any time after receiving the first dose of TAK-981 during the DLT assessment period (Cycle 1) or who received all planned TAK-981 doses and 1 administration of pembrolizumab in Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: TAK-981 40 mg | Dose Escalation: TAK-981 60 mg | Dose Escalation: TAK-981 90 mg | Dose Escalation: TAK-981 120 mg
Number analyzed (Participants) | 3 | 6 | 30 | 19
Participants | 0 | 0 | 2 | 1

3. Primary Outcome: Phase 1: Number of Participants With Grade 3 or Higher Treatment Emergent Adverse Events (TEAEs)
Description: AE means any untoward medical occurrence in a participant administered a pharmaceutical product. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product whether or not it is related to the medicinal product. A TEAE was defined as an adverse event which occurred on or after the first dose of study drug and no more than 30 days after the last dose of study drug. A severity grade was evaluated as per the NCI CTCAE Version 5.0, except for CRS, which was assessed by ASTCT Consensus Grading for CRS.
Time Frame: Up to approximately 24 months
Population: Safety Analysis Set included participants who received at least 1 dose, even if incomplete, of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: TAK-981 40 mg | Dose Escalation: TAK-981 60 mg | Dose Escalation: TAK-981 90 mg | Dose Escalation: TAK-981 120 mg
Number analyzed (Participants) | 3 | 6 | 33 | 19
Participants | 0 | 2 | 20 | 15

4. Primary Outcome: Phase 1: Number of Participants With One or More Serious Adverse Events (SAEs)
Description: An SAE is any untoward medical occurrence that results in death; is life-threatening; requires inpatient hospitalization or prolongation of present hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect or is a medically important event that may not be immediately life-threatening or result in death or hospitalization, but may jeopardize the participant or may require intervention to prevent one of other outcomes listed in definition above, or involves suspected transmission via a medicinal product of an infectious agent.
Time Frame: Up to approximately 24 months
Population: Safety Analysis Set included participants who received at least 1 dose, even if incomplete, of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: TAK-981 40 mg | Dose Escalation: TAK-981 60 mg | Dose Escalation: TAK-981 90 mg | Dose Escalation: TAK-981 120 mg
Number analyzed (Participants) | 3 | 6 | 33 | 19
Participants | 0 | 3 | 17 | 10

5. Primary Outcome: Phase 1: Number of Participants With One or More TEAEs Leading to Dose Modifications and Treatment Discontinuation
Description: An AE is any untoward medical occurrence in a participant administered a medicinal investigational drug. The untoward medical occurrence does not necessarily have to have a causal relationship with treatment. A TEAE is defined as an AE that occurs after administration of first dose of study drug and through 30 days after last dose of study drug or until start of subsequent antineoplastic therapy.
Time Frame: Up to approximately 24 months
Population: Safety Analysis Set included participants who received at least 1 dose, even if incomplete, of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: TAK-981 40 mg | Dose Escalation: TAK-981 60 mg | Dose Escalation: TAK-981 90 mg | Dose Escalation: TAK-981 120 mg
Number analyzed (Participants) | 3 | 6 | 33 | 19
Participants
  TEAE Resulting in Dose Modifications of TAK-981 | 0 | 3 | 22 | 11
  TEAE Resulting in Dose Modifications of Pembrolizumab | 0 | 3 | 15 | 4
  TEAE Resulting in Drug Discontinuation of TAK-981 | 0 | 1 | 3 | 2
  TEAE Resulting in Drug Discontinuation of Pembrolizumab | 0 | 1 | 4 | 1

6. Primary Outcome: Phase 1: Number of Participants With Clinically Significant Laboratory Values
Description: Laboratory parameters included clinical chemistry, hematology, and urinalysis. Participants with at least 1 Grade 3 or 4 Lab Abnormalities were reported.
Time Frame: Up to approximately 24 months
Population: Safety Analysis Set included participants who received at least 1 dose, even if incomplete, of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: TAK-981 40 mg | Dose Escalation: TAK-981 60 mg | Dose Escalation: TAK-981 90 mg | Dose Escalation: TAK-981 120 mg
Number analyzed (Participants) | 3 | 6 | 33 | 19
Participants
  Hematology | 1 | 3 | 7 | 6
  Serum Chemistry | 1 | 1 | 7 | 5
  Coagulation | 0 | 0 | 0 | 1

7. Primary Outcome: Phase 2: Overall Response Rate (ORR) as Assessed by the Investigator According to RECIST, Version 1.1
Description: ORR is defined as the percentage of participants who achieve Complete Response (CR) and Partial Response (PR) (determined by the investigator) during the study according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
Time Frame: Up to approximately 25 months
Population: Response-Evaluable Analysis Set included participants who had received at least 1 dose of study drug, had sites of measurable disease at baseline, and 1 postbaseline disease assessment, or were discontinued due to symptomatic deterioration or death before a postbaseline evaluation happened.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 90 mg | Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 120 mg | Dose Expansion: Cohort B: Cervical Cancer TAK-981 90 mg | Dose Expansion: Cohort C: MSS-CRC TAK-981 90 mg | Dose Expansion: Cohort D: Cutaneous Melanoma TAK-981 90 mg | Dose Expansion: Cohort E: Squamous NSCLC TAK-981 90 mg | Dose Expansion: Cohort F: CPI Refractory Squamous and Non-squamous NSCLC TAK-981 90 mg
Number analyzed (Participants) | 10 | 8 | 20 | 9 | 28 | 13 | 4
percentage of participants | 20 [2.52 to 55.61] | 0 [0.00 to 36.94] | 30 [11.89 to 54.28] | 0 [0.00 to 33.63] | 25 [10.69 to 44.87] | 7.7 [0.19 to 36.03] | 0 [0.00 to 60.24]

8. Secondary Outcome: Phase 1: Cmax: Maximum Observed Plasma Concentration for TAK-981
Time Frame: Cycle 1 (each cycle is 21 days) Days 1 and 8 pre-dose and at multiple timepoints (up to 24 hours)
Population: Pharmacokinetic (PK) Analysis Set included participants with sufficient dosing and PK data to reliably estimate 1 or more PK parameters. Number of participants analyzed is the number of participants available for analysis during the specified time-point.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/ml)
Arm/Group | Dose Escalation: TAK-981 40 mg | Dose Escalation: TAK-981 60 mg | Dose Escalation: TAK-981 90 mg | Dose Escalation: TAK-981 120 mg
Number analyzed (Participants) | 3 | 6 | 33 | 19
nanograms per milliliter (ng/ml)
  Cycle 1 Day 1 | 335 (282) | 728 (396) | 888 (423) | 1290 (571)
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 6 | 30 | 17
  Cycle 1 Day 8 | 280 (167) | 448 (206) | 780 (524) | 1270 (770)

9. Secondary Outcome: Phase 1: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-981
Time Frame: Cycle 1 (each cycle is 21 days) Days 1 and 8 pre-dose and at multiple timepoints (up to 24 hours)
Population: PK Analysis Set included participants with sufficient dosing and PK data to reliably estimate 1 or more PK parameters. Number of participants analyzed is the number of participants available for analysis during the specified time-point.
Measure: Median (Full Range); unit: hours
Arm/Group | Dose Escalation: TAK-981 40 mg | Dose Escalation: TAK-981 60 mg | Dose Escalation: TAK-981 90 mg | Dose Escalation: TAK-981 120 mg
Number analyzed (Participants) | 3 | 6 | 33 | 19
hours
  Cycle 1 Day 1 | 1.22 [1.20 to 1.23] | 1.27 [1.00 to 1.47] | 1.17 [1.00 to 1.88] | 1.20 [1.00 to 1.72]
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 6 | 30 | 17
  Cycle 1 Day 8 | 1.18 [1.17 to 1.25] | 1.41 [1.00 to 1.70] | 1.22 [1.00 to 3.10] | 1.28 [0.98 to 1.50]

10. Secondary Outcome: Phase 1: AUC0-t: Area Under the Plasma Concentration-time Curve From Time 0 to Time t Over the Dosing Interval for TAK-981
Time Frame: Cycle 1 (each cycle is 21 days) Days 1 and 8 pre-dose and at multiple timepoints (up to 24 hours)
Population: PK Analysis Set included participants with sufficient dosing and PK data to reliably estimate 1 or more PK parameters. Overall number of participants analyzed is the number of participants with data available for analysis. Number of participants analyzed is the number of participants available for analysis during the specified time-point.
Measure: Mean (Standard Deviation); unit: hours*ng/mL
Arm/Group | Dose Escalation: TAK-981 40 mg | Dose Escalation: TAK-981 60 mg | Dose Escalation: TAK-981 90 mg | Dose Escalation: TAK-981 120 mg
Number analyzed (Participants) | 3 | 6 | 32 | 18
hours*ng/mL
  Cycle 1 Day 1 | 880 (427) | 1370 (517) | 1950 (735) | 2580 (949)
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 5 | 28 | 16
  Cycle 1 Day 8 | 814 (290) | 976 (232) | 1780 (908) | 2640 (1260)

11. Secondary Outcome: Phase 1: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-981
Time Frame: Cycle 1 (each cycle is 21 days) Days 1 and 8 pre-dose and at multiple timepoints (up to 24 hours)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: hours*ng/mL
Arm/Group | Dose Escalation: TAK-981 40 mg | Dose Escalation: TAK-981 60 mg | Dose Escalation: TAK-981 90 mg | Dose Escalation: TAK-981 120 mg
Number analyzed (Participants) | 3 | 6 | 32 | 17
hours*ng/mL
  Cycle 1 Day 1 | 909 (432) | 1400 (530) | 2020 (760) | 2660 (1020)
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 5 | 27 | 16
  Cycle 1 Day 8 | 845 (292) | 1010 (233) | 1830 (942) | 2750 (1320)

12. Secondary Outcome: Phase 1: t1/2z: Terminal Disposition Phase Half-life for TAK-981
Time Frame: Cycle 1 (each cycle is 21 days) Days 1 and 8 pre-dose and at multiple timepoints (up to 24 hours)
Population: as for outcome 10
Measure: Median (Full Range); unit: hours
Arm/Group | Dose Escalation: TAK-981 40 mg | Dose Escalation: TAK-981 60 mg | Dose Escalation: TAK-981 90 mg | Dose Escalation: TAK-981 120 mg
Number analyzed (Participants) | 3 | 6 | 32 | 17
hours
  Cycle 1 Day 1 | 5.88 [5.82 to 6.16] | 5.58 [5.04 to 6.03] | 5.72 [3.31 to 10.43] | 6.79 [5.93 to 8.14]
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 5 | 27 | 16
  Cycle 1 Day 8 | 5.83 [5.69 to 6.33] | 5.68 [5.22 to 6.44] | 6.06 [4.18 to 9.13] | 6.67 [5.26 to 8.08]

13. Secondary Outcome: Phase 1: CL: Total Clearance After Intravenous Administration for TAK-981
Time Frame: Cycle 1 (each cycle is 21 days) Days 1 and 8 pre-dose and at multiple timepoints (up to 24 hours)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: liters per hour (L/h)
Arm/Group | Dose Escalation: TAK-981 40 mg | Dose Escalation: TAK-981 60 mg | Dose Escalation: TAK-981 90 mg | Dose Escalation: TAK-981 120 mg
Number analyzed (Participants) | 3 | 6 | 32 | 17
liters per hour (L/h)
  Cycle 1 Day 1 | 51.1 (23.2) | 47.2 (14.8) | 51.3 (19.6) | 51.0 (18.4)
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 5 | 27 | 16
  Cycle 1 Day 8 | 51.7 (19.3) | 62.5 (15.5) | 57.0 (21.8) | 53.8 (26.8)

14. Secondary Outcome: Phase 1: Vss: Volume of Distribution at Steady State After Intravenous Administration for TAK-981
Time Frame: Cycle 1 (each cycle is 21 days) Days 1 and 8 pre-dose and at multiple timepoints (up to 24 hours)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: liters (L)
Arm/Group | Dose Escalation: TAK-981 40 mg | Dose Escalation: TAK-981 60 mg | Dose Escalation: TAK-981 90 mg | Dose Escalation: TAK-981 120 mg
Number analyzed (Participants) | 3 | 6 | 32 | 17
liters (L)
  Cycle 1 Day 1 | 312 (203) | 181 (56.9) | 240 (115) | 240 (98.5)
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 5 | 27 | 16
  Cycle 1 Day 8 | 323 (178) | 314 (109) | 300 (129) | 271 (150)

15. Secondary Outcome: Phases 1 and 2: Disease Control Rate (DCR)
Description: DCR is defined as the percentage of participants who achieved stable disease (SD) or better (CR + PR + SD determined by the investigator) >6 weeks during the trial in the response-evaluable population.
Time Frame: Phase 1: Up to approximately 24 months, Phase 2: Up to approximately 25 months
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 120 mg: Participants with non-squamous NSCLC received TAK-981 as IV infusion on Days 1, 4, 8 and 11 or Days 1 and 8 in each 21-day Treatment Cycle up to disease progression or 24-months and pembrolizumab 200 mg IV infusion as a fixed dose every 3 weeks on Day 1 of 21-day Treatment Cycle for a maximum of 24 months.
Arm/Group | Dose Escalation: TAK-981 40 mg | Dose Escalation: TAK-981 60 mg | Dose Escalation: TAK-981 90 mg | Dose Escalation: TAK-981 120 mg | Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 90 mg | Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 120 mg | Dose Expansion: Cohort B: Cervical Cancer TAK-981 90 mg | Dose Expansion: Cohort C: MSS-CRC TAK-981 90 mg | Dose Expansion: Cohort D: Cutaneous Melanoma TAK-981 90 mg | Dose Expansion: Cohort E: Squamous NSCLC TAK-981 90 mg | Dose Expansion: Cohort F: CPI Refractory Squamous and Non-squamous NSCLC TAK-981 90 mg
Number analyzed (Participants) | 3 | 6 | 33 | 18 | 10 | 8 | 20 | 9 | 28 | 13 | 4
percentage of participants | 33.3 [0.84 to 90.57] | 50.0 [11.81 to 88.19] | 30.3 [15.59 to 48.71] | 44.4 [21.53 to 69.24] | 80.0 [44.39 to 97.48] | 62.5 [24.49 to 91.48] | 55.0 [31.53 to 76.94] | 22.2 [2.81 to 60.01] | 67.9 [47.65 to 84.12] | 30.8 [9.09 to 61.43] | 0 [0.00 to 60.24]

16. Secondary Outcome: Phases 1 and 2: Durable Response Rate (DRR)
Description: DRR is defined as the rate of objective responses (CR + PR) maintained for at least 6 months initiating at any time within 12 months of commencing therapy.
Time Frame: Phase 1: Up to approximately 24 months, Phase 2: Up to approximately 25 months
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Escalation: TAK-981 40 mg | Dose Escalation: TAK-981 60 mg | Dose Escalation: TAK-981 90 mg | Dose Escalation: TAK-981 120 mg | Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 90 mg | Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 120 mg | Dose Expansion: Cohort B: Cervical Cancer TAK-981 90 mg | Dose Expansion: Cohort C: MSS-CRC TAK-981 90 mg | Dose Expansion: Cohort D: Cutaneous Melanoma TAK-981 90 mg | Dose Expansion: Cohort E: Squamous NSCLC TAK-981 90 mg | Dose Expansion: Cohort F: CPI Refractory Squamous and Non-squamous NSCLC TAK-981 90 mg
Number analyzed (Participants) | 3 | 6 | 33 | 18 | 10 | 8 | 20 | 9 | 28 | 13 | 4
percentage of participants | 0 [0.00 to 70.76] | 16.7 [0.42 to 64.12] | 6.1 [0.74 to 20.23] | 0 [0.00 to 18.53] | 10.0 [0.25 to 44.50] | 0 [0.00 to 36.94] | 0 [0.00 to 16.84] | 0 [0.00 to 33.63] | 10.7 [2.27 to 28.23] | 0 [0.00 to 24.71] | 0 [0.00 to 60.24]

17. Secondary Outcome: Phases 1 and 2: Duration of Response (DOR)
Description: DOR is defined as a time from the time of first documentation of tumor response to the first recorded occurrence of disease progression (PD) or death from any cause (whichever occurs first), through end of study.
Time Frame: Phase 1: Up to approximately 24 months, Phase 2: Up to approximately 25 months
Population: Response-Evaluable Analysis Set included participants who had received at least 1 dose of study drug, had sites of measurable disease at baseline, and 1 postbaseline disease assessment, or were discontinued due to symptomatic deterioration or death before a postbaseline evaluation happened. Overall number of participants analyzed is the number of participants with events.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Dose Escalation: TAK-981 40 mg | Dose Escalation: TAK-981 60 mg | Dose Escalation: TAK-981 90 mg | Dose Escalation: TAK-981 120 mg | Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 90 mg | Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 120 mg | Dose Expansion: Cohort B: Cervical Cancer TAK-981 90 mg | Dose Expansion: Cohort C: MSS-CRC TAK-981 90 mg | Dose Expansion: Cohort D: Cutaneous Melanoma TAK-981 90 mg | Dose Expansion: Cohort E: Squamous NSCLC TAK-981 90 mg | Dose Expansion: Cohort F: CPI Refractory Squamous and Non-squamous NSCLC TAK-981 90 mg
Number analyzed (Participants) | 0 | 1 | 3 | 1 | 1 | 0 | 2 | 0 | 3 | 1 | 0
hours |  | 17.12 [NA to NA] — Lower and upper limit of 95% Confidence Interval was not estimable for a single participant. | 7.39 [4.17 to NA] — Upper limit of 95% Confidence Interval was not estimable due to censoring. | 3.71 [NA to NA] — Lower and upper limit of 95% Confidence Interval was not estimable for a single participant. | 7.62 [NA to NA] — Lower and upper limit of 95% Confidence Interval was not estimable for a single participant. |  | NA [4.67 to NA] — Median and upper limit of 95% Confidence Interval was not estimable due to censoring. |  | NA [7.26 to NA] — Median and upper limit of 95% Confidence Interval was not estimable due to censoring. | 4.34 [NA to NA] — Lower and upper limit of 95% Confidence Interval was not estimable for a single participant. |

18. Secondary Outcome: Phases 1 and 2: Progression-free Survival (PFS)
Description: PFS is defined as time from the date of the first dose administration to the date of first documentation of PD or death due to any cause whichever occurs first, through the end of the study.
Time Frame: Phase 1: Up to approximately 24 months, Phase 2: Up to approximately 25 months
Population: as for outcome 17
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Escalation: TAK-981 40 mg | Dose Escalation: TAK-981 60 mg | Dose Escalation: TAK-981 90 mg | Dose Escalation: TAK-981 120 mg | Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 90 mg | Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 120 mg | Dose Expansion: Cohort B: Cervical Cancer TAK-981 90 mg | Dose Expansion: Cohort C: MSS-CRC TAK-981 90 mg | Dose Expansion: Cohort D: Cutaneous Melanoma TAK-981 90 mg | Dose Expansion: Cohort E: Squamous NSCLC TAK-981 90 mg | Dose Expansion: Cohort F: CPI Refractory Squamous and Non-squamous NSCLC TAK-981 90 mg
Number analyzed (Participants) | 3 | 5 | 28 | 16 | 8 | 7 | 15 | 8 | 17 | 11 | 4
months | 2.00 [2.00 to NA] — Upper limit of 95% Confidence Interval was not estimable due to censoring. | 4.21 [2.00 to NA] — Upper limit of 95% Confidence Interval was not estimable due to censoring. | 1.99 [1.77 to 3.91] | 2.11 [1.41 to 6.57] | 3.71 [3.29 to 9.20] | 4.59 [1.97 to NA] — Upper limit of 95% Confidence Interval was not estimable due to censoring. | 4.14 [2.14 to 8.87] | 1.64 [1.28 to 2.00] | 8.97 [2.37 to 12.42] | 2.07 [1.87 to 2.30] | 1.28 [0.99 to NA] — Upper limit of 95% Confidence Interval was not estimable due to censoring.

19. Secondary Outcome: Phases 1 and 2: Time to Response (TTR)
Description: TTR is defined as time from the date of the first dose administration to the date of first documented PR or better.
Time Frame: Phase 1: Up to approximately 24 months, Phase 2: Up to approximately 25 months
Population: as for outcome 17
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Escalation: TAK-981 40 mg | Dose Escalation: TAK-981 60 mg | Dose Escalation: TAK-981 90 mg | Dose Escalation: TAK-981 120 mg | Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 90 mg | Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 120 mg | Dose Expansion: Cohort B: Cervical Cancer TAK-981 90 mg | Dose Expansion: Cohort C: MSS-CRC TAK-981 90 mg | Dose Expansion: Cohort D: Cutaneous Melanoma TAK-981 90 mg | Dose Expansion: Cohort E: Squamous NSCLC TAK-981 90 mg | Dose Expansion: Cohort F: CPI Refractory Squamous and Non-squamous NSCLC TAK-981 90 mg
Number analyzed (Participants) | 0 | 2 | 3 | 1 | 2 | 0 | 6 | 0 | 7 | 1 | 0
months |  | 4.17 [1.91 to NA] — Upper limit of 95% Confidence Interval was not estimable due to censoring. | NA [3.94 to NA] — Median and Upper limit of 95% Confidence Interval was not estimable due to censoring. | NA [NA to NA] — Median, lower limit and upper limit of 95% CI was not estimable due to censoring. | 4.01 [3.98 to NA] — Upper limit of 95% Confidence Interval was not estimable due to censoring. |  | 6.01 [4.04 to NA] — Upper limit of 95% Confidence Interval was not estimable due to censoring. |  | NA [NA to NA] — Median, lower limit and upper limit of 95% CI was not estimable due to censoring. | NA [NA to NA] — Median, lower limit and upper limit of 95% CI was not estimable due to censoring. |

20. Secondary Outcome: Phases 1 and 2: Time to Progression (TTP)
Description: TTP is defined as the from the date of the first dose administration to the date of the first documentation of PD as defined by standard disease criteria.
Time Frame: Phase 1: Up to approximately 24 months, Phase 2: Up to approximately 25 months
Population: as for outcome 17
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Escalation: TAK-981 40 mg | Dose Escalation: TAK-981 60 mg | Dose Escalation: TAK-981 90 mg | Dose Escalation: TAK-981 120 mg | Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 90 mg | Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 120 mg | Dose Expansion: Cohort B: Cervical Cancer TAK-981 90 mg | Dose Expansion: Cohort C: MSS-CRC TAK-981 90 mg | Dose Expansion: Cohort D: Cutaneous Melanoma TAK-981 90 mg | Dose Expansion: Cohort E: Squamous NSCLC TAK-981 90 mg | Dose Expansion: Cohort F: CPI Refractory Squamous and Non-squamous NSCLC TAK-981 90 mg
Number analyzed (Participants) | 3 | 5 | 25 | 15 | 8 | 6 | 13 | 6 | 14 | 11 | 4
months | 2.00 [2.00 to NA] — Upper limit of 95% Confidence Interval was not estimable due to censoring. | 4.21 [2.00 to NA] — Upper limit of 95% Confidence Interval was not estimable due to censoring. | 2.07 [1.87 to 4.04] | 2.07 [1.41 to 6.93] | 3.71 [3.29 to 9.20] | 4.01 [1.97 to NA] — Upper limit of 95% Confidence Interval was not estimable due to censoring. | 5.34 [2.20 to 8.87] | 1.76 [1.28 to NA] — Upper limit of 95% Confidence Interval was not estimable due to censoring. | 9.17 [4.11 to NA] — Upper limit of 95% Confidence Interval was not estimable due to censoring. | 2.07 [1.87 to 2.30] | 1.28 [0.99 to NA] — Upper limit of 95% Confidence Interval was not estimable due to censoring.

21. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: OS is defined as the time from the date of the first dose administration to the date of death. Participants without documentation of death at the time of analysis were censored at the date last known to be alive.
Time Frame: Up to approximately 25 months
Population: as for outcome 17
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 90 mg | Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 120 mg | Dose Expansion: Cohort B: Cervical Cancer TAK-981 90 mg | Dose Expansion: Cohort C: MSS-CRC TAK-981 90 mg | Dose Expansion: Cohort D: Cutaneous Melanoma TAK-981 90 mg | Dose Expansion: Cohort E: Squamous NSCLC TAK-981 90 mg | Dose Expansion: Cohort F: CPI Refractory Squamous and Non-squamous NSCLC TAK-981 90 mg
Number analyzed (Participants) | 1 | 4 | 9 | 2 | 8 | 1 | 1
months | NA [NA to NA] — Median, Lower limit and Upper limit of 95% CI was not estimable due to censoring. | 10.12 [5.16 to NA] — Upper limit of 95% Confidence Interval was not estimable due to censoring. | 14.55 [5.42 to NA] — Upper limit of 95% Confidence Interval was not estimable due to censoring. | NA [4.21 to NA] — Median and Upper limit of 95% CI was not estimable due to censoring. | NA [11.43 to NA] — Median and Upper limit of 95% CI was not estimable due to censoring. | NA [NA to NA] — Median and Upper limit of 95% CI was not estimable due to censoring. | NA [1.28 to NA] — Median and Upper limit of 95% CI was not estimable due to censoring.

22. Secondary Outcome: Fold Change From Baseline in TAK-981-/Small Ubiquitin-like Modifier (SUMO) Adduct Formation in Peripheral Blood Lymphocytes
Description: The level of TAK-981-SUMO adduct formation was evaluated by flow cytometry as the percentage of adduct formed in peripheral blood lymphocytes. Fold change from baseline was calculated as: Post-treatment value / Baseline value. Positive change denotes improvement.
Time Frame: Cycle 1 Day 1 (1 hour, 4 hours, 8 hours) and Day 8 (Pre-dose, 1 hour, 4 hours and 8 hours) (Cycle length = 21 days)
Population: Pharmacodynamic Analysis Set included participants who provided evaluable blood samples (Cycle 1, Day 1 predose sample and at least 1 postdose sample). Overall number of participants analyzed is the number of participants with data available for analysis. Number of participants analyzed is the number of participants available for analysis during the specified time-point.
Measure: Mean (Standard Deviation); unit: unitless ratio
Arm/Group | Dose Escalation: TAK-981 40 mg | Dose Escalation: TAK-981 60 mg | Dose Escalation: TAK-981 90 mg | Dose Escalation: TAK-981 120 mg
Number analyzed (Participants) | 3 | 6 | 18 | 13
unitless ratio
  Cycle 1 Day 1: 1 Hour Post Dose | 8.1 (1.06) | 7.0 (3.12) | 8.5 (3.38) | 8.4 (2.40)
  Cycle 1 Day 1: 4 Hours Post Dose | 5.1 (0.82) | 5.0 (1.90) | 6.0 (1.80) | 6.3 (1.70)
  Cycle 1 Day 1: 6-8 Hours Post Dose | 4.6 (0.61) | 4.5 (1.87) | 5.3 (1.58) | 5.5 (1.29)
  Cycle 1 Day 8: Predose: number analyzed (Participants) | 3 | 6 | 16 | 12
  Cycle 1 Day 8: Predose | 3.5 (0.53) | 2.6 (0.96) | 2.7 (1.43) | 2.0 (0.68)
  Cycle 1 Day 8: 1 Hour Post Dose: number analyzed (Participants) | 3 | 6 | 16 | 10
  Cycle 1 Day 8: 1 Hour Post Dose | 11.9 (3.52) | 7.7 (2.88) | 9.2 (4.68) | 8.7 (2.01)
  Cycle 1 Day 8: 4 Hours Post Dose: number analyzed (Participants) | 3 | 6 | 14 | 11
  Cycle 1 Day 8: 4 Hours Post Dose | 7.5 (1.52) | 6.0 (2.66) | 6.4 (2.90) | 6.1 (2.12)
  Cycle 1 Day 8: 6-8 Hours Post Dose: number analyzed (Participants) | 3 | 6 | 14 | 11
  Cycle 1 Day 8: 6-8 Hours Post Dose | 6.5 (1.08) | 5.1 (2.30) | 5.7 (2.64) | 5.6 (1.96)

23. Secondary Outcome: Fold Change From Baseline in SUMO 2/3 Inhibition in Peripheral Blood Lymphocytes
Description: SUMO pathway inhibition in blood was evaluated by flow cytometry in peripheral blood lymphocytes with an antibody recognizing SUMO 2/3 chains. Fold change from baseline was calculated as: Post-treatment value / Baseline value.
Time Frame: Cycle 1 Day 1 (1 hour, 4 hours, 8 hours) and Day 8 (Pre-dose, 1 hour, 4 hours and 8 hours) (Cycle length = 21 days)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: unitless ratio
Arm/Group | Dose Escalation: TAK-981 40 mg | Dose Escalation: TAK-981 60 mg | Dose Escalation: TAK-981 90 mg | Dose Escalation: TAK-981 120 mg
Number analyzed (Participants) | 3 | 6 | 18 | 13
unitless ratio
  Cycle 1 Day 1: 1 Hour Post Dose | 0.7 (0.14) | 0.6 (0.21) | 0.6 (0.18) | 0.5 (0.08)
  Cycle 1 Day 1: 4 Hours Post Dose | 0.8 (0.07) | 0.6 (0.12) | 0.9 (0.54) | 0.6 (0.11)
  Cycle 1 Day 1: 6-8 Hours Post Dose | 0.8 (0.08) | 0.7 (0.19) | 1.0 (0.68) | 0.7 (0.34)
  Cycle 1 Day 8: Predose: number analyzed (Participants) | 3 | 6 | 16 | 12
  Cycle 1 Day 8: Predose | 0.9 (0.24) | 1.0 (0.35) | 0.9 (0.36) | 0.7 (0.39)
  Cycle 1 Day 8: 1 Hour Post Dose: number analyzed (Participants) | 3 | 6 | 16 | 10
  Cycle 1 Day 8: 1 Hour Post Dose | 0.6 (0.14) | 0.6 (0.23) | 0.7 (0.34) | 0.4 (0.15)
  Cycle 1 Day 8: 4 Hours Post Dose: number analyzed (Participants) | 3 | 6 | 14 | 11
  Cycle 1 Day 8: 4 Hours Post Dose | 0.7 (0.22) | 0.6 (0.15) | 0.8 (0.58) | 0.5 (0.17)
  Cycle 1 Day 8: 6-8 Hours Post Dose: number analyzed (Participants) | 3 | 6 | 14 | 11
  Cycle 1 Day 8: 6-8 Hours Post Dose | 0.7 (0.29) | 0.6 (0.11) | 0.9 (0.53) | 0.6 (0.22)

24. Secondary Outcome: Phase 2: Percentage of Participants With One or More Treatment Emergent Adverse Events (TEAEs)
Description: An AE is any untoward medical occurrence in a participant administered a medicinal investigational drug. The untoward medical occurrence does not necessarily have to have a causal relationship with treatment. A TEAE is defined as an AE that occurs after administration of first dose of study drug and through 30 days after last dose of study drug or until start of subsequent antineoplastic therapy. AEs were evaluated according to NCI CTCAE, Version 5.0 except CRS, which was graded according to ASTCT Consensus Grading for CRS.
Time Frame: Up to approximately 25 months
Population: Safety Analysis Set included participants who received at least 1 dose, even if incomplete, of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 90 mg | Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 120 mg | Dose Expansion: Cohort B: Cervical Cancer TAK-981 90 mg | Dose Expansion: Cohort C: MSS-CRC TAK-981 90 mg | Dose Expansion: Cohort D: Cutaneous Melanoma TAK-981 90 mg | Dose Expansion: Cohort E: Squamous NSCLC TAK-981 90 mg | Dose Expansion: Cohort F: CPI Refractory Squamous and Non-squamous NSCLC TAK-981 90 mg
Number analyzed (Participants) | 14 | 9 | 21 | 9 | 28 | 15 | 4
percentage of participants | 100 | 100 | 100 | 100 | 100 | 93.3 | 100

25. Secondary Outcome: Phase 2: Number of Participants With Grade 3 or Higher Treatment Emergent Adverse Events (TEAEs)
Description: An AE means any untoward medical occurrence in a participant administered a pharmaceutical product. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product whether or not it is related to the medicinal product. A TEAE was defined as an adverse event which occurred on or after the first dose of study drug and no more than 30 days after the last dose of study drug. A severity grade was evaluated as per the NCI CTCAE Version 5.0, except for CRS, which was assessed by ASTCT Consensus Grading for CRS.
Time Frame: Up to approximately 25 months
Population: Safety Analysis Set included participants who received at least 1 dose, even if incomplete, of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 90 mg | Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 120 mg | Dose Expansion: Cohort B: Cervical Cancer TAK-981 90 mg | Dose Expansion: Cohort C: MSS-CRC TAK-981 90 mg | Dose Expansion: Cohort D: Cutaneous Melanoma TAK-981 90 mg | Dose Expansion: Cohort E: Squamous NSCLC TAK-981 90 mg | Dose Expansion: Cohort F: CPI Refractory Squamous and Non-squamous NSCLC TAK-981 90 mg
Number analyzed (Participants) | 14 | 9 | 21 | 9 | 28 | 15 | 4
Participants | 7 | 5 | 18 | 8 | 14 | 4 | 2

26. Secondary Outcome: Phase 2: Number of Participants With One or More TEAEs Leading to Dose Modifications and Treatment Discontinuation
Description: as for outcome 5
Time Frame: Up to approximately 25 months
Population: Safety Analysis Set included participants who received at least 1 dose, even if incomplete, of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 90 mg | Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 120 mg | Dose Expansion: Cohort B: Cervical Cancer TAK-981 90 mg | Dose Expansion: Cohort C: MSS-CRC TAK-981 90 mg | Dose Expansion: Cohort D: Cutaneous Melanoma TAK-981 90 mg | Dose Expansion: Cohort E: Squamous NSCLC TAK-981 90 mg | Dose Expansion: Cohort F: CPI Refractory Squamous and Non-squamous NSCLC TAK-981 90 mg
Number analyzed (Participants) | 14 | 9 | 21 | 9 | 28 | 15 | 4
Participants
  TEAE Resulting in Dose Modifications of TAK-981 | 11 | 6 | 15 | 5 | 15 | 6 | 4
  TEAE Resulting in Dose Modifications of Pembrolizumab | 7 | 5 | 12 | 4 | 13 | 2 | 4
  TEAE Resulting in Drug Discontinuation of TAK-981 | 1 | 1 | 6 | 0 | 6 | 1 | 0
  TEAE Resulting in Drug Discontinuation of Pembrolizumab | 1 | 3 | 4 | 0 | 3 | 1 | 0

ADVERSE EVENTS:
Time Frame: Phase 1: Up to approximately 24 months, Phase 2: Up to approximately 25 months
Description: Safety Analysis Set included participants who received at least 1 dose, even if incomplete, of study drug.
Groups:
- Dose Escalation: TAK-981 120 mg: Participants received TAK-981, 120 mg, IV infusion, on Days 1, 4, 8 and 11 or Days 1 and 8 in each 21-day Treatment Cycle and pembrolizumab 200 mg, IV infusion, as a fixed dose every 3 weeks on Day 1 of 21-day Treatment Cycle until the RP2D was determined (for a maximum of 24 months).
- Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 120 mg: Participants with non-squamous NSCLC received TAK-981 120 mg as IV infusion on Days 1, 4, 8 and 11 or Days 1 and 8 in each 21-day Treatment Cycle up to disease progression or 24-months and pembrolizumab 200 mg IV infusion as a fixed dose every 3 weeks on Day 1 of 21-day Treatment Cycle for a maximum of 24 months.
- Dose Expansion: Cohort F: CPI Refractory Squamous or Non-squamous NSCLC TAK-981 90 mg: Participants with CPI refractory squamous or non-squamous NSCLC received TAK-981 90 mg as IV infusion on Days 1, 4, 8 and 11 or Days 1 and 8 in each 21-day Treatment Cycle up to disease progression or 24-months and pembrolizumab 200 mg IV infusion as a fixed dose every 3 weeks on Day 1 of 21-day Treatment Cycle for a maximum of 24 months.
Arm/Group | Dose Escalation: TAK-981 40 mg | Dose Escalation: TAK-981 60 mg | Dose Escalation: TAK-981 90 mg | Dose Escalation: TAK-981 120 mg | Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 90 mg | Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 120 mg | Dose Expansion: Cohort B: Cervical Cancer TAK-981 90 mg | Dose Expansion: Cohort C: MSS-CRC TAK-981 90 mg | Dose Expansion: Cohort D: Cutaneous Melanoma TAK-981 90 mg | Dose Expansion: Cohort E: Squamous NSCLC TAK-981 90 mg | Dose Expansion: Cohort F: CPI Refractory Squamous or Non-squamous NSCLC TAK-981 90 mg
All-Cause Mortality (participants affected / at risk) | 2/3 | 2/6 | 8/33 | 4/19 | 2/14 | 4/9 | 9/21 | 2/9 | 8/28 | 2/15 | 1/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 3/6 | 17/33 | 10/19 | 3/14 | 4/9 | 11/21 | 4/9 | 14/28 | 5/15 | 3/4
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 33/33 | 19/19 | 14/14 | 9/9 | 21/21 | 9/9 | 28/28 | 14/15 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation: TAK-981 40 mg (N=3) | Dose Escalation: TAK-981 60 mg (N=6) | Dose Escalation: TAK-981 90 mg (N=33) | Dose Escalation: TAK-981 120 mg (N=19) | Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 90 mg (N=14) | Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 120 mg (N=9) | Dose Expansion: Cohort B: Cervical Cancer TAK-981 90 mg (N=21) | Dose Expansion: Cohort C: MSS-CRC TAK-981 90 mg (N=9) | Dose Expansion: Cohort D: Cutaneous Melanoma TAK-981 90 mg (N=28) | Dose Expansion: Cohort E: Squamous NSCLC TAK-981 90 mg (N=15) | Dose Expansion: Cohort F: CPI Refractory Squamous or Non-squamous NSCLC TAK-981 90 mg (N=4)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aortic aneurysm rupture (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aplasia pure red cell (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 3 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related thrombosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Orchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transfusion-related acute lung injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation: TAK-981 40 mg (N=3) | Dose Escalation: TAK-981 60 mg (N=6) | Dose Escalation: TAK-981 90 mg (N=33) | Dose Escalation: TAK-981 120 mg (N=19) | Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 90 mg (N=14) | Dose Expansion: Cohort A: Non-squamous NSCLC TAK-981 120 mg (N=9) | Dose Expansion: Cohort B: Cervical Cancer TAK-981 90 mg (N=21) | Dose Expansion: Cohort C: MSS-CRC TAK-981 90 mg (N=9) | Dose Expansion: Cohort D: Cutaneous Melanoma TAK-981 90 mg (N=28) | Dose Expansion: Cohort E: Squamous NSCLC TAK-981 90 mg (N=15) | Dose Expansion: Cohort F: CPI Refractory Squamous or Non-squamous NSCLC TAK-981 90 mg (N=4)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1 | 1 | 5 | 0 | 0 | 0 | 0
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 3 | 1 | 3 | 0 | 1
Abnormal weight gain (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 7 | 1 | 4 | 2 | 4 | 0 | 2 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 16 | 6 | 3 | 2 | 13 | 3 | 7 | 2 | 2
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angular cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 5 | 3 | 4 | 1 | 4 | 2 | 5 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 13 | 2 | 4 | 4 | 4 | 2 | 3 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 2 | 0 | 0 | 3 | 4 | 0 | 1 | 3 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 1 | 3 | 0 | 0 | 0 | 2 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Balanitis candida (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 5 | 0 | 2 | 1 | 4 | 1 | 1 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 3 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
CD4 lymphocytes decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 1 | 2 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 12 | 11 | 5 | 2 | 1 | 1 | 4 | 1 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 3 | 1 | 0 | 0 | 3 | 1 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 4 | 2 | 0 | 3 | 2 | 10 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 3 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 10 | 6 | 1 | 4 | 4 | 3 | 5 | 1 | 3
Defaecation urgency (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dengue fever (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 4 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 9 | 9 | 3 | 2 | 7 | 3 | 7 | 3 | 1
Diplopia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 3 | 1 | 2 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 5 | 4 | 2 | 1 | 2 | 1 | 1 | 0 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Electrocardiogram ST-T segment abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epididymal cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 13 | 4 | 5 | 5 | 6 | 5 | 9 | 0 | 1
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 6 | 4 | 3 | 0 | 2 | 2 | 5 | 0 | 0
Herpes simplex reactivation (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 2 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 2 | 2 | 1 | 0 | 3 | 2 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 3 | 5 | 0 | 2 | 1 | 1 | 0 | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 1 | 1 | 2 | 1 | 1 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 3 | 2 | 1 | 0 | 1 | 1 | 2 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 5 | 0 | 2 | 0 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 7 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Infusion site extravasation (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 2 | 0 | 1 | 1 | 2 | 1 | 1 | 1 | 0
Interleukin level increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intestinal polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lip oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 4 | 0 | 3 | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 4 | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 1 | 0 | 3 | 0 | 5 | 0 | 0
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 8 | 5 | 3 | 6 | 9 | 2 | 13 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Nervous system neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 4 | 1 | 2 | 0 | 2 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 2 | 3 | 2 | 2 | 2 | 0 | 5 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 3 | 2 | 2 | 2 | 1 | 0 | 0 | 1
Orchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paroxysmal arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Penile oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 6 | 3 | 1 | 0 | 0 | 0 | 2 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 2 | 1 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Poor peripheral circulation (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procalcitonin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 1 | 1 | 2 | 0 | 6 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulpitis dental (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 17 | 14 | 9 | 4 | 11 | 3 | 11 | 6 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 4 | 1 | 0 | 3 | 0 | 3 | 0 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin candida (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Steroid diabetes (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 8 | 8 | 4 | 2 | 1 | 3 | 8 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Swelling face (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
T-lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 4 | 2 | 1 | 1 | 1 | 2 | 1 | 1
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 0
Urethritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 4 | 1 | 1 | 1 | 6 | 1 | 5 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 7 | 5 | 4 | 2 | 5 | 2 | 4 | 1 | 1
Weight decreased (Investigations) | 0 | 0 | 2 | 2 | 0 | 1 | 2 | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-06-22): https://cdn.clinicaltrials.gov/large-docs/50/NCT04381650/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-08): https://cdn.clinicaltrials.gov/large-docs/50/NCT04381650/SAP_001.pdf